CLINICAL TRIAL: NCT04002687
Title: A Randomized, Double-blind, Placebo Controlled Parallel Group Study in Heathy Adult Subjects to Determine the Tolerability and Safety of Atovaquone-proguanil (ATV-PG) Co-administered With Amodiaquine (AQ)
Brief Title: Determine the Tolerability and Safety of Atovaquone-proguanil (ATV-PG) Co-administered With Amodiaquine (AQ)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APM/18/1702001
Record Dates: First submitted 2019-06-17; First posted 2019-06-28 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Fifty-two subjects will be enrolled and randomized to one of the four treatment (Cohorts 1 to 4) in a ratio of 4:3:3:3 as described below:
  * Treatment 1 (n=16) - ATV-PG 1000-400 mg + AQ 612 mg;
  * Treatment 2 (n=12) - ATV-PG 1000-400 mg + AQ unmatched placebo;
  * Treatment 3 (n=12) - ATV-PG unmatched placebo + AQ 612 mg;
  * Treatment 4 (n=12) - ATV-PG unmatched placebo + AQ unmatched placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be conducted in a double-blind fashion whereby subjects and clinical study site staff are blinded. Because the placebo tablets are not an exact match for the active treatment, tablets will be administered by an un-blinded member of clinical study staff, who will protect the blinding from both subjects and all other site staff. Dosing will take place behind a curtain and during IMP administration the subjects will be blindfolded. The pharmacy staff preparing the investigational products will not be blinded to study drug assignment. During the study, the individual randomisation codes will be kept in the site's clinical trials pharmacy, accessible to the pharmacy personnel only. Upon completion of the study, after the database lock and after the blind is revealed, the randomisation list will be filed in the Trial Master File. Sponsor staff involved in clinical decision-making (such as those involved in SRC decisions) will be blinded to study drug assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ATV-PG 1000-400 mg + AQ 612 mg (Experimental): T1 (n=16) - Atovaquone (ATV),Proguanil (PG) 1000-400 mg + Amodiaquine (AQ) 612 mg on days 1,2, 3.
  Interventions: Drug: ATV-PG 1000-400 mg + AQ 612 mg
- ATV-PG 1000-400 mg + AQ unmatched placebo (Active Comparator): T 2 (n=12) - Atovaquone (ATV)-Proguanil (PG) 1000-400 mg + Amodiaquine (AQ) unmatched placebo on days 1,2, 3.
  Interventions: Drug: ATV-PG 1000-400 mg + AQ 612 mg
- ATV-PG unmatched placebo + AQ 612 mg (Active Comparator): T 3 (n=12) - Atovaquone (ATV)-Proguanil (PG) unmatched placebo + Amodiaquine (AQ) 612 mg on days 1,2, 3.
  Interventions: Drug: ATV-PG 1000-400 mg + AQ 612 mg
- ATV-PG unmatched placebo + AQ unmatched placebo (Placebo Comparator): T 4 (n=12) - Atovaquone (ATV)-Proguanil (PG) unmatched placebo + AQ unmatched placebo on days 1,2, 3.
  Interventions: Drug: ATV-PG 1000-400 mg + AQ 612 mg

INTERVENTIONS:
Drug: ATV-PG 1000-400 mg + AQ 612 mg — The dosing will be carried out by an unblinded member of the investigator's staff. Dosing will take place behind a curtain and during IMP administration the subjects will be blindfolded. ATV-PG (or placebo) will always be given first, then AQ (or placebo).
  Other Names: ATV-PG 1000-400 mg + AQ unmatched placebo; ATV-PG unmatched placebo + AQ 612 mg

SUMMARY:
The aim of the study is to determine the tolerability and safety of ATV-PG + AQ, ATV-PG + AQ placebo, ATV-PG placebo + AQ, and ATV-PG placebo + AQ placebo administered once daily for 3 days to healthy adult male and female subjects.This study in healthy adults is the first step towards establishing the tolerability and safety of the approved doses of ATV-PG and AQ when co-administered. If considered acceptable based on the findings of this study, the tolerability, safety and PE will subsequently be assessed, within the target geographical areas.

DETAILED DESCRIPTION:
Although the tolerability and safety of ATV-PG and AQ alone are well established, additive tolerability signals are possible on co-administration. Four treatment arms will be used: ATV-PG + AQ placebo, ATV-PG placebo + AQ, ATV-PG placebo + AQ placebo, as well as ATV-PG + AQ. This will facilitate discrimination of the contribution of the treatments to any tolerability signal. In the event that ATV-PG + AQ is not considered sufficiently well tolerated, data on the individual agents will provide an indication of whether ATV-PG or AQ are suitable partner drugs for other combinations.

Thus, this study will evaluate in healthy adults, whether the tolerability and safety profile of once daily administration of ATV-PG + AQ for 3 days supports future use in Seasonal Malaria Chemoprevention (SMC), which will entail administration on a monthly basis to an apparently healthy population of children of 3 months of age and older, for the duration of the malaria season.

This study will also determine the pharmacokinetics of ATV, PG, CG (active metabolite of PG), AQ and DEAQ (active metabolite of AQ).

Given the ultimate target population (children in Southern and Easter Africa in areas in which SMC with SPAQ is not currently deployed due to SP resistance), the study will be carried out in healthy subjects of sub-Saharan African origin (defined as subjects whose parents were both born in sub-Saharan Africa).

ELIGIBILITY:
Inclusion Criteria:

1) Male or female, of sub-Saharan African origin (both parents born in sub-Saharan Africa), aged ≥18 to ≤45 years at the date of signing informed consent which is defined as the beginning of the Screening Period.

2. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to follow the following contraception requirements. Contraception must start one complete menstrual cycle prior to the first day of dosing and continue until at least 90 days after the end of the systemic exposure of the study drug (90 days after the last study drug administration).

Female subjects who are documented as being of non-childbearing potential are exempt from contraception requirements. Documentation of non-childbearing potential must include at least one of the following criteria:

* Postmenopausal - evidence of menopause based on a combination of amenorrhea for at least one year and increased serum follicle-stimulating hormone (FSH) level (> 30 IU/L), or
* Surgical sterilization - evidence of hysterectomy and/or bilateral oophorectomy.

All female subjects of childbearing potential and all male subjects with female partnersof childbearing potential, who are pregnant or breastfeeding must practice highly effective or acceptable methods of contraception (defined below) when having heterosexual intercourse.

Sexual abstinence, defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug treatment can be considered a highly effective method of contraception for female and male subjects. Reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the subject.

Contraception methods for female subjects in this study:

* Hormonal contraception:

  * Combined i.e. oestrogen- and progestogen-containing (oral, intravaginal or transdermal)
  * Progestogen-only (oral, injectable or implantable)
  * Intrauterine hormone-releasing system (IUS)
* Intrauterine device (IUD) or
* Bilateral tubal occlusion
* Male partner vasectomised (with documented evidence of azoospermia if possible)
* (Male partner uses) male condom with or without spermicide
* Cap, diaphragm, or sponge with spermicide

Contraception methods for male subjects in this study:

* Male condom with or without spermicide
* Vasectomy (with documented evidence of azoospermia if possible) 3. Subjects must agree not to donate sperm or ova from the time of the first administration of study medication until 3 months after the end of the systemic exposure of the study drugs. 4. Subjects must have a body weight of at least 50 kg and a body mass index (BMI) between 18-25.0 kg/m² inclusive at screening.

  5. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation (haematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with the subject's participation in or ability to complete the study as assessed by the Investigator.

  6. Ability to swallow 8 capsules/tablets at a time or consecutively. 7. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (R2) (2016) and applicable regulations, before completing any study-related procedures.

  8. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. Current or recurrent disease (e.g., cardiovascular, haematological, neurological,endocrine, immunological, renal, hepatic or gastrointestinal or other conditions) that could affect the action, absorption, or disposition of ATV-PG or AQ, or could affect clinical assessments or clinical laboratory evaluations.
2. Any significant history of seizures or epilepsy.
3. Current or relevant history of physical or psychiatric illness that may require treatment or make the subject unlikely to fully comply with the requirements or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
4. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study may influence the result of the study, or the subject's ability to participate in the study.
5. Documented retinopathy.
6. History of photosensitivity.
7. History of malaria.
8. Subjects have travelled to malaria endemic regions for more than a total of 4 weeks within the past 12 months (as per Global Malaria Risk: https://www.malariasite.com/malaria-risk/ [20]-)
9. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.
10. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QTc interval changes. This includes subjects with any of the following (at screening or Day -1):

    * Sinus node dysfunction.
    * Clinically significant PR (PQ) interval prolongation.
    * Intermittent second or third degree AV block.
    * Complete bundle branch block.
    * Sustained cardiac arrhythmia's including (but not limited to) atrial fibrillation or supraventricular tachycardia; any symptomatic arrhythmia with the exception of isolated extra systoles.
    * Abnormal T wave morphology which may impact on the QT/QTc assessment.
    * QT interval corrected using the Fridericia's formula (QTcF) > 450 ms (males and females).
    * Any other ECG abnormalities in the standard 12-lead ECG and 24-hour 12 lead Holter ECG or an equivalent assessment which in the opinion of the Investigator will interfere with the ECG analysis.

    Subjects with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the PI.
11. Has vital signs outside of the following normal range at screening or Day -1:

    1. Blood pressure (BP):

Supine BP (after at least 5 minutes of supine rest):

* Systolic blood pressure: 90 - 140 mmHg.
* Systolic blood pressure drop of >20mmHg on standing (at screening only)
* Diastolic blood pressure: 40 - 90 mmHg. b. Pulse rate (after at least 5 minutes of supine rest):
* Less than 40 or greater than 100 beats per minute 12. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening; 13.

  1. AST, ALT or bilirubin measurement above the laboratory reference ranges, at screening or Day -1.
  2. Haemoglobin or platelet count outside of the laboratory reference ranges.
  3. or any other clinically significant abnormal haematological measurement (per the Investigator's discretion). 14. Positive test results for alcohol or drugs of abuse at screening or Day -1. 15. Female subjects who are pregnant (including a positive serum pregnancy test at screening and on Day-1) or breastfeeding.

     16. History or clinical evidence of substance and/or alcohol abuse within the 2 years before screening. Alcohol abuse is defined as regular weekly intake of more than 14 units (for both males and females), using the following NHS alcohol tracker http://www.nhs.uk/Tools/Pages/drinks-tracker.aspx. 17. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, electronic cigarettes) within 3 months prior to the planned first day of dosing.

     18. Has used any other prescription medication (excluding hormonal contraception, hormone replacement therapy) within 14 days or 10 half-lives (whichever is longer) prior to Day 1 of the dosing period that the Investigator judges is likely to interfere with the study or pose an additional risk in participating.

     19. Has used any over-the-counter medication (including multivitamin, herbal, or homeopathic preparations; excluding paracetamol - up to 1g paracetamol per day permitted) during the 7 days or 5 half-lives of the drug (whichever is longer) prior to Day 1 of the dosing period, that the Investigator judges is likely to interfere with the study or pose an additional risk in participating.

     20. Has used any medication listed on the Flockhart table (http://medicine.iupui.edu/clinpharm/ddis/main-table/) that is either a moderate or strong inhibitor or inducer of CYP450 within 30 days or 5 half-lives (whichever is longer) prior to the planned first day of dosing.

     21. Has received an investigational product or been treated with an investigational device within 90 days or 5 half-lives (whichever is the longer) prior to first drug administration.

     22. Known or suspected intolerance or hypersensitivity to the investigational product, atovaquone, proguanil or amodiaquine, any closely related compound, or any of the stated ingredients.

     23. History of significant allergic reaction (anaphylaxis, angioedema) to any product (food, pharmaceutical, etc).

     24. Has donated or lost 400 mL blood (excluding plasma) or more within the last 16 weeks preceding the first day of dosing.

     25. Has a mental incapacity or language barriers precluding adequate understanding, cooperation, and compliance with the study requirements 26. An inability to follow a standardised diet and meal schedule or inability to fast, as required during the study.

     27. Subjects have veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins that are difficult to locate access or puncture veins with a tendency to rupture during or after puncture).

     28. Prior screen failure (where the cause of the screen failure is not deemed to be temporary), randomisation, participation, or enrolment in this study. Subjects who initially failed due to temporary non-medically significant issues are eligible for rescreening once the cause has resolved.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) will be assessed of the approved dose of ATV-PG and the adult equivalent of the approved SMC dose of AQ when administered alone and in combination and in combination, in comparison with placebo. | Day 1 to Day 29 post dose, (Day 36 +/- 1 day including follow up)
  TEAEs will include clinical signs, nausea, vomiting and diarrhea, proportion of subjects with clinically relevant changes in laboratory safety tests (hematology, chemistry (in particular ALT, AST and bilirubin increases) and urinalysis), proportion of subjects with morphological and/or rhythm abnormalities on electrocardiogram (ECG), proportion of subjects with clinically significant changes in ECG time intervals (PR, QRS, QT and QTc intervals) and proportion of subjects with clinically significant changes in vital signs (systolic blood pressure, diastolic blood pressure and pulse rate).

SECONDARY OUTCOMES:
To measure the the maximum observed plasma concentration (Cmax) of atovaquone (ATV), proguanil (PG) and cycloguanil (CG), and amodiaquine (AQ) and desethyl-amodiaquine (DEAQ) following administration of ATV-PG and AQ alone and in combination. | Day 1 to Day 22
  To measure the maximum observed plasma concentration (Cmax).
To measure the maximum plasma concentration (tmax) of atovaquone (ATV), proguanil (PG) and cycloguanil (CG), and amodiaquine (AQ) and desethyl-amodiaquine (DEAQ) following administration of ATV-PG and AQ alone and in combination. | Day 1 to Day 22
  To measure time the maximum plasma concentration (tmax).
To measure the area under the plasma concentration-time curve from time zero to last detectable plasma concentration (AUC0-t) of atovaquone, proguanil and cycloguanil, and amodiaquine and desethyl-amodiaquine (DEAQ) following administration. | Day 1 to Day 22
  To measure the area under the plasma concentration-time curve from time to zero to last detectable plasmaconcentration (AUC0-t).
To measure the area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf) of atovaquone (ATV), proguanil (PG) and cycloguanil (CG), and amodiaquine (AQ) and desethyl-amodiaquine (DEAQ) following administr | Day 1 to Day 22
  To measure the area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf)
To measure the terminal elimination rate constant (λz) of atovaquone (ATV), proguanil (PG) and cycloguanil (CG), and amodiaquine (AQ) and desethyl-amodiaquine (DEAQ) following administr | Day 1 to Day 22
  To measure the terminal elimination rate constant (λz).
To measure the terminal elimination half-life (t1/2) of atovaquone (ATV), proguanil (PG) and cycloguanil (CG), and amodiaquine (AQ) and desethyl-amodiaquine (DEAQ) following administr | Day 1 to Day 22
  To measure the terminal elimination half-life (t1/2).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD FRCA FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd., Croydon, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De- Identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months after study completion.
Access Criteria: Requestors will be required to sign a Data Access Agreement.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT04002687/SAP_000.pdf
  • Study Protocol (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04002687/Prot_001.pdf